CLINICAL TRIAL: NCT00130416
Title: Improving Chronic Disease Care With PatientSite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 51757
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Depression; Pain; Mobility Difficulty
Keywords: behavior; randomized trial; communication; patient; internet; coaching; self-efficacy; nurse; primary care; physician; screening; survey; pain; mobility; disability; depression
MeSH Terms: conditions — Depression; Pain; Behavior; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: E-mail coaching to improve patient communication with doctor

SUMMARY:
The overall goal of this randomized, controlled trial is to test whether educational interventions - directed toward empowering patients and delivered via the Beth Israel Deaconess Medical Center (BIDMC's) secure patient Internet portal PatientSite - can improve the outcomes and satisfaction with care of adult primary care patients with 3 common conditions: chronic pain, depression, and progressive difficulty walking.

DETAILED DESCRIPTION:
PURPOSE OF PROTOCOL:

The overall goal of this randomized, controlled trial is to test whether educational interventions - directed toward empowering patients and delivered via the BIDMC's secure patient Internet portal PatientSite - can improve outcomes and satisfaction with care of adult primary care patients with 3 common conditions: chronic pain, depression, and progressive difficulty walking.

Primary study outcomes include improvement among intervention patients in:

1. detection and treatment of the target conditions;
2. patient-reported signs and symptoms of pain, depression, and impaired lower extremity mobility;
3. patient-reported quality of life, patient-clinician communication, and satisfaction with care; and
4. health care utilization. The secondary outcome is physicians' views that the intervention improved the efficiency and quality of care they deliver.

The specific aims of the project are:

1. to improve physicians' detection and treatment of patient-reported pain, depression, and impaired walking among intervention patients compared to controls;
2. to reduce patient-reported symptoms of chronic pain, depression, and impaired walking among intervention patients compared to controls;
3. to improve patient-reported quality of life, patient-clinician communication, and satisfaction with care among intervention patients compared to controls; and 4. to improve physicians' assessments of the efficiency of office visits and quality of care they provided for the 3 study conditions.

SIGNIFICANCE AND BACKGROUND FOR THE STUDY:

Chronic conditions affect 99 million Americans and limit the daily lives of 41 million (Institute for Health & Aging 1996). Moreover, these conditions are often unrecognized. Myriad reasons contribute to the under-diagnosis of chronic conditions, including problems with patient-clinician communication, providers' lack of awareness of the prevalence of these conditions or how to screen for them, and abbreviated office visits (e.g., Beckman 1999). Many conditions are difficult to ascertain, such as depression and pain, without objective and readily apparent indicators of impairment. Some persons believe that mobility difficulties are an inevitable consequence of aging, and something that physicians can do little to help, and primary care physicians generally have little formal training in mobility assessments (Iezzoni 2003a). An accurate, timely, and inexpensive way to identify and address chronic conditions could potentially transform the care of patients, enhance their quality of life, improve clinicians' work life, and mitigate the social cost of these conditions.

This project will test whether a secure patient Internet portal is a useful conduit for information that can improve patient care, by screening patients for certain conditions, communicating the results directly to the patient and their physician, empowering patients to address these condition with their physicians, facilitating clinicians' actions, and activating patients to participate in their own care.

PATIENTSITE:

PatientSite is a secure, personalized messaging system serving BIDMC and affiliated sites. It allows patients to communicate confidentially with their physicians and the physicians' staff via the Web. Patients are eligible to enroll in PatientSite if one of their physicians has agreed to use PatientSite. Data in PatientSite are encrypted and password protected. Patients register online, and receive passwords from administrators at their own practice site in order to confirm the patient's identity. Patients and clinicians must use a confidential password to obtain access to the system. To alert PatientSite users to the presence of a message, PatientSite sends users a traditional email message that they have a PatientSite message, along with a link to the PatientSite Web portal.

DESCRIPTION OF RESEARCH PROTOCOL:

The researchers are conducting a randomized, controlled trial of a PatientSite intervention designed to improve pain, depression, and impaired mobility among primary care patients, among other outcomes.

The researchers are recruiting physicians who currently use PatientSite from among those practicing at BIDMC's academic primary care practice and at 2 community practices affiliated with BIDMC. Patients of physicians who agree to participate are potentially eligible for the study. Two weeks before their next scheduled primary care office visit, The researchers are sending these patients an e-mail invitation via PatientSite to participate in the study. The e-mail briefly describes the study (including the procedures for randomization) and links patients to a complete, electronic informed consent form as well as standard HIPAA disclosures.

Patients who electronically sign the informed consent, thereby agreeing to participate in the study, are sent a screening questionnaire asking about signs and symptoms of chronic pain, depression, and difficulty walking. Persons who screen positive for at least one of these three conditions are enrolled in the study and randomized to intervention and control groups.

Patients randomized to the intervention electronically receive an e-mail message containing additional information about ways to address the condition during their primary care visit within the upcoming two weeks. The message includes condition-specific suggestions about how to discuss the problem with their clinician, along with standard tips about communicating with doctors. It provides a confidential link to an "electronic advocate" - a clinical nurse "e-Coach" who coaches (advises) the patient online about how to address the problem with their physician in the upcoming appointment.

Patients randomized to the control group receive an e-mail containing links to federal government Web sites containing general health information unrelated to the target conditions.

The researchers are surveying both intervention and control group subjects via PatientSite 1 week and 3 months after their index visit to find out about their visit and their satisfaction with care, their clinical outcomes relating to the target conditions, and use of additional health care services. At one week post-visit, the researchers are specifically asking whether they discussed the condition with their clinician and whether the clinician did anything about it. The researchers are further asking patients who did not address the symptom with their physician for the reason. Three months after the index visit, the researchers re-administer the screening instruments used at baseline in order to ascertain change in the target conditions, quality of life, health communication, and satisfaction. The researchers also review patients' medical records to abstract demographic information (age, gender, race, ethnicity, primary language), administrative data (insurance type, utilization of health services), and clinical characteristics (from the index visit note written by the physician) to corroborate discussion and management of target conditions, and to assess medical care utilization.

The researchers are surveying participating physicians at the conclusion of the study to obtain their perceptions about the impact of the intervention on their work including time burdens and quality of care. In addition, the researchers are reviewing the electronic medical records to ascertain provider and utilization outcome information at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patients aged 18 and older, of participating physicians within 5 internal medicine practices in Boston
* Registered users of patient-provider internet portal called PatientSite
* Screened positive for depression, chronic pain, or lower extremity mobility difficulty

Exclusion Criteria:

* Current treatment for screened condition by medical or surgical specialist or other appropriate licensed health professional such as a physical therapist or mental health counselor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 2004-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Resolution or improvement in screened chronic condition
Improved communication with primary care doctor
Improved patient satisfaction
Improved physician satisfaction

SECONDARY OUTCOMES:
Favorable clinician assessment of the impact of the screening intervention on the efficiency and quality of care they deliver

CONTACTS AND LOCATIONS:
Overall Officials: Lisa I Iezzoni, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Leveille SG, Huang A, Tsai SB, Allen M, Weingart SN, Iezzoni LI. Health coaching via an internet portal for primary care patients with chronic conditions: a randomized controlled trial. Med Care. 2009 Jan;47(1):41-7. doi: 10.1097/MLR.0b013e3181844dd0. PMID 19106729
- See also: Website for patient-doctor internet portal — https://www.patientsite.org/
- See also: website for Health e-Technologies Initiative, a national program office of the Robert Wood Johnson Foundation — http://www.hetinitiative.org/